CLINICAL TRIAL: NCT05248620
Title: Prophylactic Antibiotic Treatment in End Stage Kidney Disease and Central Venous Catheter as Hemodialysis Vascular Access
Brief Title: Prophylactic Antibiotic Treatment in Hemodialysis
Acronym: PANTHEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-20026735
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis
Keywords: Blood stream infections; Severe culture negative infections; Central venous catheter; Prophylactic antibiotics

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, single-blinded, placebo controlled study, with blinded endpoint evaluation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Amoxicillin/placebo is provided in identical containers. Amoxicillin and placebo tablets are looking similar, but by decision of the Danish Medicines Agency amoxicillin tablets must not be removed from the original folio packing prior to use. Clindamycin active and placebo tablets look similar (incapsulated), and are provided in identical containers. Study medicine will be provided by 1-2 nurses at each site, who are unblinded. The patients and care providers are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Amoxicillin/clavulanic acid 500/125mg, tablets, will be administered before each hemodialysis for 6 months
  Interventions: Drug: Amoxicillin Clavulanic 500/125mg or placebo
- Placebo (Placebo Comparator): Placebo tablets, similar to the active drug, will be administered before each hemodialysis for 6 months
  Interventions: Drug: Amoxicillin Clavulanic 500/125mg or placebo

INTERVENTIONS:
Drug: Amoxicillin Clavulanic 500/125mg or placebo — Prophylactic antibiotic treatment
  Other Names: Aurobindo

SUMMARY:
The purpose of this study is to assess the efficacy of prophylactic antibiotic treatment on blood stream infections and severe culture negative infections, in patients on newly started hemodialysis(HD), with a central venous catheter as vascular access.

DETAILED DESCRIPTION:
After being informed about the study and potential risks all eligible patients, giving written informed consent will be included in the study. At week 0 patients will be randomized in a single blinded manner (participants and care providers) in a 1:1 manner to receive 500/125mg amoxicillin/clavulanic acid 30-120 minutes before each hemodialysis with a central venous catheter (CVC) as vascular access, or corresponding placebo. The timing of antibiotic administration has been established in a pilot-study in order to secure a sufficient concentration of antibiotics during the dialysis session. In case of side effects to amoxicillin/clavulanic acid, the prophylactic antibiotic will be shifted to 600mg clindamycin. Total treatment period with prophylactic antibiotics is 6 months, with a 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Kidney Disease (ESKD) patients who receive an uncuffed or cuffed CVC for expected chronic HD, regardless of previous ESKD treatment modality (PD or KTX) and hemodialysis access (AV-fistula or AV-graft))
* ≥18 years
* Ability to understand the study background, risk and benefit of treatment and to give written informed consent

Exclusion Criteria:

* Unable to give informed consent
* Known intolerance to beta-lactam antibiotics and clindamycin
* Active infection treated with antibiotics
* Breastfeeding
* Pregnancy. In women of childbearing age, an approved birth control must be ensured at least 1 month before and during all the 6 months of antibiotic/placebo treatment.

Patients may be rescreened later i.e. within a time period of one month from start of HD, if exclusion criteria are reversible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Blood stream infection (BSI) | ≤ 6 months after randomization
  Hospitalization for BSI
Number of patients with Severe blood culture negative infection | ≤ 6 months after randomization
  Hospitalization ≥ 3 days due to infection defined as: C-reactive protein (CRP) ≥ 75 and negative blood cultures, treated with iv antibiotics

SECONDARY OUTCOMES:
Number of patients with BSI or severe blood culture negative infection | ≤ 6 months after randomization
  Each of the components in the primary endpoint
Mortality | ≤ 6 months after randomization
  All-cause mortality

OTHER OUTCOMES:
Number of patients with Sepsis | ≤ 6 months after randomization
  Hospitalization due to sepsis or septic shock
Number of patients with Deep tissue infection | ≤ 6 months after randomization
  Infective endocarditis, osteomyelitis, and spondylodiscitis
Number of patients with Autoinfection | ≤ 6 months after randomization
  Frequency of BSI autoinfection
Number of patients with Clostridium difficile infection | ≤ 6 months after randomization
  Clostridium difficile infection - numbers and days of admission
Mortality due to infection - number of patients | ≤ 6 months after randomization
  Mortality due to infection
Number of CVC removals | ≤ 6 months after randomization
  CVC removal due to CVC infection
Use of Antibiotics in Difined Daily Doses | ≤ 6 months after randomization
  Total use of antibiotics in Defined Daily Doses
Healt-care economics | ≤ 6 months after randomization
  Health-care related economic consequences due to hospitalization and treatment of the disease
Number of patients with Extended Spectrum Beta-Lactamase (ESBL) infection | ≤ 6 months after randomization
  ESBL infections - number of patients and days of admission
Number of patients with Methicillin-resistant Staphylococcus aureus (MRSA) infection | ≤ 6 months after randomization
  MRSA infections - number of patients and days of admission
Number of patients with Carbapenemase-Producing Organisms (CPO) infection | ≤ 6 months after randomization
  CPO infections - number og patients and days of admission
Number of patients with Vancomycin-resistant enterococci (VRE) infection | ≤ 6 months after randomization
  VRE infections - number of patients and days of admission
Number of patients with Cardiovascular events | ≤ 6 months after randomization
  Hospitalization with acute myocardial infarction, worsening heart failure or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Niels E Bruun, Professor, Principal Investigator — Dept. cardiology, Zealand University Hospital, Roskilde, Denmark
Locations (7):
- Denmark (7):
  - Rigshospitalet, Copenhagen, Capital Region
  - Herlev-Gentofte Hospital, Copenhagen, Capital Region
  - North Zealand Hospital Hillerød, Hillerød, Capital Region
  - Aarhus University Hospital, Aarhus, Middle Region
  - Aalborg University Hospital, Aalborg, North Region
  - ZUH Roskilde, Roskilde, Region Sjælland
  - Odense University Hospital, Odense, Region South

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Gupta V, Yassin MH. Infection and hemodialysis access: an updated review. Infect Disord Drug Targets. 2013 Jun;13(3):196-205. doi: 10.2174/1871526511313030008. PMID 24001331
- [Background] Vogelzang JL, van Stralen KJ, Noordzij M, Diez JA, Carrero JJ, Couchoud C, Dekker FW, Finne P, Fouque D, Heaf JG, Hoitsma A, Leivestad T, de Meester J, Metcalfe W, Palsson R, Postorino M, Ravani P, Vanholder R, Wallner M, Wanner C, Groothoff JW, Jager KJ. Mortality from infections and malignancies in patients treated with renal replacement therapy: data from the ERA-EDTA registry. Nephrol Dial Transplant. 2015 Jun;30(6):1028-37. doi: 10.1093/ndt/gfv007. Epub 2015 Jan 29. PMID 25637641
- [Background] Aslam S, Vaida F, Ritter M, Mehta RL. Systematic review and meta-analysis on management of hemodialysis catheter-related bacteremia. J Am Soc Nephrol. 2014 Dec;25(12):2927-41. doi: 10.1681/ASN.2013091009. Epub 2014 May 22. PMID 24854263
- [Background] Sarnak MJ, Jaber BL. Mortality caused by sepsis in patients with end-stage renal disease compared with the general population. Kidney Int. 2000 Oct;58(4):1758-64. doi: 10.1111/j.1523-1755.2000.00337.x. PMID 11012910
- [Background] Jaber BL. Bacterial infections in hemodialysis patients: pathogenesis and prevention. Kidney Int. 2005 Jun;67(6):2508-19. doi: 10.1111/j.1523-1755.2005.00364.x. No abstract available. PMID 15882306
- [Background] de Jager DJ, Grootendorst DC, Jager KJ, van Dijk PC, Tomas LM, Ansell D, Collart F, Finne P, Heaf JG, De Meester J, Wetzels JF, Rosendaal FR, Dekker FW. Cardiovascular and noncardiovascular mortality among patients starting dialysis. JAMA. 2009 Oct 28;302(16):1782-9. doi: 10.1001/jama.2009.1488. PMID 19861670
- [Background] Chaudry MS, Gislason GH, Kamper AL, Rix M, Dahl A, Ostergaard L, Fosbol EL, Lauridsen TK, Oestergaard LB, Hassager C, Torp-Pedersen C, Bruun NE. The impact of hemodialysis on mortality risk and cause of death in Staphylococcus aureus endocarditis. BMC Nephrol. 2018 Sep 3;19(1):216. doi: 10.1186/s12882-018-1016-0. PMID 30176809
- [Background] Chaudry MS, Carlson N, Gislason GH, Kamper AL, Rix M, Fowler VG Jr, Torp-Pedersen C, Bruun NE. Risk of Infective Endocarditis in Patients with End Stage Renal Disease. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1814-1822. doi: 10.2215/CJN.02320317. Epub 2017 Oct 3. PMID 28974524
- [Background] Nelveg-Kristensen KE, Laier GH, Heaf JG. Risk of death after first-time blood stream infection in incident dialysis patients with specific consideration on vascular access and comorbidity. BMC Infect Dis. 2018 Dec 20;18(1):688. doi: 10.1186/s12879-018-3594-7. PMID 30572826
- [Background] Sakhuja A, Nanchal RS, Gupta S, Amer H, Kumar G, Albright RC, Kashani KB. Trends and Outcomes of Severe Sepsis in Patients on Maintenance Dialysis. Am J Nephrol. 2016;43(2):97-103. doi: 10.1159/000444684. Epub 2016 Mar 10. PMID 26959243